CLINICAL TRIAL: NCT05561088
Title: A Single-center, Prospective, Randomized, Controlled Study of Mechanical Thrombectomy Followed by Acupuncture for Acute Ischemic Stroke
Brief Title: Efficacy and Safety of Head Acupuncture After Mechanical Thrombectomy for Acute Ischemic Stroke
Acronym: HEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sy-11-2022-124
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Acupuncture; Acute Ischemic Stroke; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Mechanical thrombectomy was followed by acupuncture and guideline-based conventional treatment
  Interventions: Other: Scalp Acupuncture; Other: The treatment recommended in the guidelines for acute ischemic stroke was administered
- control group (Experimental): Conventional treatment based on guidelines was administered after mechanical thrombectomy
  Interventions: Other: The treatment recommended in the guidelines for acute ischemic stroke was administered

INTERVENTIONS:
Other: Scalp Acupuncture — mplementation plan of head needle: The middle frontal line (MS1), the middle parietal line (MS5) and the back parietal and temporal oblique line (MS7) in the International Standardization Program for the Name of the first needle Point in 1989 were selected, and the needles were inserted along the shape of each section. One needle was inserted into the middle frontal line and the middle parietal line, and two needles were inserted into the back parietal and temporal oblique line. The KWD-808I pulse electrotherapy instrument produced by Changzhou Wujin Great Wall Medical Equipment Co., Ltd. is used on the needle handle after lifting, inserting and twisting. The continuous waveform was used, the voltage was 2-4 V, the frequency was 60-80 times /min, the intensity was tolerated by the patient, the needle was kept for 30min, and the treatment was performed once a day.
  Arms: experimental group
Other: The treatment recommended in the guidelines for acute ischemic stroke was administered — The treatment recommended in the guidelines for acute ischemic stroke was administered

SUMMARY:
To evaluate the efficacy and safety of head acupuncture combined with endovascular therapy for cerebral infarction compared with endovascular therapy alone

DETAILED DESCRIPTION:
Control group: Mechanical thrombectomy followed by the guideline recommended treatment for acute ischemic stroke;

Experimental group: After mechanical thrombectomy, head acupuncture and the treatment regimen recommended by the guideline for acute ischemic stroke were administered

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Patients with acute ischemic stroke who received endovascular treatment within 24 hours of onset;
* 6 < NIHSS ≤25;
* ASPECT score ≥6 points;
* Signed Informed consent.

Exclusion Criteria:

* CT or brain MRI confirmed intracranial tumor and intracranial hemorrhage;
* Contraindications of contrast media;
* Dementia or mental illness，unable to cooperate with treatment and follow-up;
* The expected survival time was less than 3 months;
* Women who are pregnant, planning to become pregnant or breastfeeding;
* Currently participating in other clinical trials.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of Modified rankin scale (mRS) score ≤2 | 90 days after onset
  The modified rankin Scale (mRS) score ≤2 indicates that the patient has the ability to live independently.

SECONDARY OUTCOMES:
National Institute of Health stroke scale(NIHSS) score | 10 days after onset
  NIHSS scores range from 0 to 42, with higher scores indicating more severe nerve damage.
Modified rankin scale (mRS) score | 90 days after onset
  Modified rankin scale (mRS) Score is used to measure the neurological function recovery status of patients after stroke, and its score ranges from 0 to 6
Incidence of cerebral hemorrhage | 7 days after randomization
  No hemorrhage was found on the first head CT/MRI after cerebral infarction, but intracranial hemorrhage was found on the second head CT/MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Xi 'an No.3 Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No